CLINICAL TRIAL: NCT04827394
Title: Preventing Hypothermia in Moderate and Late Preterm Neonates - a Pilot Randomized Controlled Trial
Brief Title: Neonatal Warming to Prevent Hypothermia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12752
Record Dates: First submitted 2021-03-04; First posted 2021-04-01 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Intervention Model Description: 1:1 using a block randomization scheme stratified by gestational age
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention group (Experimental): In the intervention group, the infant will be placed on the thermal mattress, then wrapped.
  Interventions: Device: Neonatal warming mattress; Device: Sterile polyethylene wrap
- Control group (No Intervention): In the non-intervention group, the infant will be delivered onto the sterile field as per standard of care.

INTERVENTIONS:
Device: Neonatal warming mattress — Babies will be warmed with a standard neonatal transport warming mattress immediately after birth.
  Arms: Intervention group
Device: Sterile polyethylene wrap — Babies will be wrapped in a sterile polyethylene wrap prior to arrival at the warmer.
  Arms: Intervention group

SUMMARY:
Researchers are proposing a pilot randomized controlled trial evaluating the benefit of immediately warming preterm babies using a warming mattress and a plastic wrap, while delaying clamping the umbilical cord at the time of c-section in babies born between 32 and 36 weeks to determine if it reduces the risk of hypothermia.

DETAILED DESCRIPTION:
The trial will be advertised and introduced to patients admitted to the OU Children's Hospital labor and delivery or antepartum units by research nurses. Interested participants will be consented. Researchers are choosing to only include patients undergoing non-emergent cesarean in order to improve their ability to control parameters such as room temperature and labor-related clinical or subclinical maternal infection, which are known confounders. Further, they are limiting their investigation to fetuses 32-36 weeks gestation, since this population represents the largest preterm delivery population. Recruitment and randomization will be stratified by gestational age with an aim to enroll at least 44 pregnancies at 32-34 weeks and 6 days and 20 pregnancies between 35-36 weeks and 6 days. Last, it is impossible to recruit patients outside of the inpatient setting for a study investigating preterm delivery, as such deliveries are rarely predictable in the outpatient setting. There will only be one site for this study, the OU Children's Hospital labor and delivery and antepartum units.

The proposed study is a pragmatic randomized controlled pilot trial of neonatal warming techniques with participants allocated in a 1:1 ratio using a random block allocation table using blocks of size 4 and 6 that are stratified by gestational age ranges of 35-36 weeks and 6 days and 32-34 weeks and 6 days. Since there cannot be a placebo intervention, neither the patient nor the neonatal team will be blinded to the group assignment. The group assignments will be made and coded by a third party at the time of randomization. Patients will be randomized to their respective groups immediately prior to surgery.

The surgical technician will be provided with the necessary neonatal wraps and mattresses in a sterile fashion, and they will ensure these are available on the surgical field once the cesarean has begun. In the intervention group, the thermal mattress will be activated immediately prior to hysterotomy and placed on the sterile field with delivery of the infant directly onto the mattress. The infant will be dried, stimulated and bulb suctioned as deemed necessary per standard of care followed by wrapping. In the non-intervention group, the infant will be delivered onto the sterile field, dried and suctioned as deemed necessary per OU standard. Cord clamping will be delayed for 60 seconds in all infants under the supervision of both the obstetrician and the neonatal resuscitation team. If either team believes delayed cord clamping is no longer considered safe, as is usual protocol, the cord will be clamped and cut and the baby will be handed off to the neonatology team. After the infant is handed to the neonatology team along with all group assignment specific materials (neonatal wrap and thermal mattress, if in the intervention group), neonatal temperature will be assessed immediately upon arrival to the resuscitation warmer using a digital thermometer placed in the axillary space. Infant temperature will be recorded at 1) arrival to the warmer, 2) after the neonatologist deems that in-room resuscitation is complete and 3) at admission to the Neonatal Intensive Care Unit (NICU), Mother Baby Unit (MBU) or Post-Anesthesia Care Unit (PACU) depending on the baby's needs; determined by the resuscitating physicians. These measurements will be recorded by research nurses in a data collection sheet. Further, the research nurse will record the time from delivery to the time it takes for the infant to arrive at the warmer. Upon arrival at the warmer, the mattress and wrap will be removed as neonatal evaluation takes place.

As immediate neonatal temperature is not generally discussed with patients unless there is an issue such as concern for infection, neonatal temperature will not be routinely discussed with all participants. Only if there is concern for neonatal infection or if there is hyperthermia (>37.5 degrees C) will the study results be discussed with the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have non-emergent cesarean deliveries (defined as at least 2 hours prior to planned cesarean)
* Gestational age between 32 weeks and 0 days and 36 weeks and 6 days determined per usual clinical parameters

Exclusion Criteria:

* Fetal anomalies or death
* Maternal diabetes
* Neonates with blistering skin conditions
* Reversed end diastolic umbilical artery flow
* Placental abruption
* Chorioamnionitis
* Monochorionic multifetal pregnancies
* Inability to provide consent
* Provider perception that patient is in significant pain and provider perceived contraindications to delayed cord clamping.

Max Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Birju Shah, MD, Principal Investigator — University of Oklahoma HSC
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share data

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The values reported reflect the total number of unique participants (mothers) assigned to each Arm.
Groups:
- Warming Mattress and Sterile Polyethylene Wrap Group: In the intervention group, the infant was placed on the thermal mattress, then wrapped.
  Neonatal warming mattress: Babies will be warmed with a standard neonatal transport warming mattress immediately after birth.
  Sterile polyethylene wrap: Babies will be wrapped in a sterile polyethylene wrap prior to arrival at the warmer.
- Standard of Care Group: In the non-intervention group, the infant will be delivered onto the sterile field as per standard of care.
Period: Overall Study
Arm/Group | Warming Mattress and Sterile Polyethylene Wrap Group | Standard of Care Group
Started | 25 | 27
Completed | 25 | 25
Not Completed | 0 | 2
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Due to the nature of the study, only females (mothers) were enrolled. The sex of the newborns was not collected.
  Participants
    Female | 25 | 25 | 50
    Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16 | 14 | 30
  Black or African American | 2 | 2 | 4
  American Indian/Alaska Native | 2 | 1 | 3
  Asian | 0 | 1 | 1
  Unknown/Not Reported | 5 | 7 | 12
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 17 | 15 | 32
  Ethnicity Unknown or Not Reported | 4 | 3 | 7
Maternal Age [Mean (Standard Deviation); unit: years] | 31.9 (6.4) | 28.7 (6.2) | 30.3 (6.3)
Gestational age [Mean (Standard Deviation); unit: days] | 241.0 (10.8) | 242.1 (11.1) | 241.6 (11.0)
Number of prenatal visits [Mean (Standard Deviation); unit: visits] | 6.5 (3.0) | 6.6 (3.3) | 6.6 (3.2)
Body Mass Index (kg/m2) [Median (Full Range); unit: kg/m2] | 34.2 [30.2 to 39.2] | 32.5 [27.9 to 40.7] | 33.35 [27.9 to 40.7]
Payor Status [Number; unit: participants]
  Private | 11 | 10 | 21
  Government/Self | 14 | 15 | 29
Recevied Prenatal Care [Number; unit: participants] | 23 | 23 | 46
Maternal Labor [Number; unit: participants] | 5 | 7 | 12
Rupture of Membranes [Number; unit: participants] | 8 | 12 | 20
Meconium Stain [Number; unit: participants] | 0 | 0 | 0
Maternal Complications [Number; unit: participants]
  Chronic Hypertension | 10 | 6 | 16
  Gestational Hypertension | 2 | 2 | 4
  Preeclampsia Without Severe Features | 0 | 3 | 3
  Preeclampsia With Severe Features | 8 | 10 | 18
  Eclampsia | 0 | 0 | 0
  HELLP | 0 | 0 | 0
  Thyroid Disorder | 0 | 2 | 2
  None | 3 | 3 | 6
NICU Admission [Number; unit: participants] | 16 | 18 | 34
Fetal Complications [Number; unit: participants]
  Twins | 3 | 3 | 6
  Fetal Growth Restriction | 1 | 4 | 5
  Oligohydramnios | 1 | 2 | 3
  Polyhydramnios | 1 | 0 | 1
  Sepsis | 1 | 1 | 2
  Death | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Temperature at Arrival to Warmer
Description: Temperature at arrival to the Warmer
Time Frame: 3 minutes
Measure: Median (Full Range); unit: degrees Celsius
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
degrees Celsius | 36.9 [36.5 to 37.3] | 37.0 [36.8 to 37.1]

2. Secondary Outcome: Temperature at Exit
Description: The temperature at exit is only available for n=21 in treatment groups and n=19 in control group.
Time Frame: 3 minutes
Measure: Median (Full Range); unit: degrees Celsius
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 21 | 19
degrees Celsius | 36.8 [36.4 to 37.0] | 36.7 [36.6 to 37.0]

3. Secondary Outcome: Temperature at NICU/Recovery
Description: Temperature at admission to NICU/Recovery
Time Frame: 24 hours
Measure: Median (Full Range); unit: degrees Celsius
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
degrees Celsius | 36.6 [36.4 to 36.8] | 36.5 [36.3 to 36.8]

4. Secondary Outcome: Peak Bilirubin
Description: Highest bilirubin level of infant based on blood test
Time Frame: Through hospital discharge up to 3 months
Measure: Median (Full Range); unit: mg/dl
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 23 | 21
mg/dl | 9.0 [5.0 to 10.0] | 9.0 [7.0 to 11.0]

5. Secondary Outcome: Duration of Respiratory Support
Description: Duration of respiratory support in the form of intubation or continuous positive airway pressure (if applicable)
Time Frame: Through hospital discharge up to 3 months
Measure: Median (Full Range); unit: hours
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 16 | 17
hours | 114.3 [2.1 to 189.9] | 31.2 [14.8 to 169.5]

6. Secondary Outcome: Length of Delayed Cord Clamp
Description: Length of delayed cord clamp in seconds
Time Frame: Up to 60 seconds after birth
Measure: Median (Full Range); unit: seconds
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
seconds | 61.0 [60.0 to 66.0] | 62.0 [33.0 to 65.0]

7. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay in days
Time Frame: Through hospital discharge up to 3 months
Measure: Median (Full Range); unit: days
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
days | 11.0 [5.0 to 20.0] | 7.0 [3.0 to 14.0]

8. Secondary Outcome: Age to Wean to Crib
Description: Age to wean to crib in days
Time Frame: Through hospital discharge up to 3 months
Measure: Median (Full Range); unit: days
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 24 | 23
days | 3.0 [0.0 to 8.0] | 1.0 [1.0 to 7.0]

9. Secondary Outcome: Hypothermia at Warmer
Description: Number of infants with hypothermia at time of arrival to warmer
Time Frame: Immediately after cord clamping (up to 60 seconds after birth)
Measure: Number; unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
participants | 6 | 2

10. Secondary Outcome: Hypothermia at Completion of Resuscitation
Description: Hypothermia at the Completion of Resuscitation
Time Frame: Through hospital discharge up to 3 months
Measure: Number; unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
participants | 6 | 3

11. Secondary Outcome: Hypothermia at NICU/Recovery
Description: Hypothermia at NICU admission /Recovery
Time Frame: Through hospital discharge up to 3 months
Measure: Number; unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
participants | 7 | 11

12. Secondary Outcome: Hyperthermia (>37.5C) at Warmer
Description: Hyperthermia (>37.5C) at arrival to Warmer
Time Frame: Through hospital discharge up to 3 months
Measure: Number; unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
participants | 2 | 1

13. Secondary Outcome: Hypoglycemia
Description: Hypoglycemia (less than 30mg/dL in the first 24 hours)
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
participants | 4 | 3

14. Secondary Outcome: Need for NICU Admission
Description: Whether or not infant was admitted to NICU
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
participants | 16 | 18

15. Secondary Outcome: Composite
Description: Composite neonatal morbidity (if applicable)
Time Frame: Through hospital discharge up to 3 months
Measure: Number; unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 25
participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Through discharge, assessed up to 3 months per participant
Description: Adverse events were collected for participants throughout their participation in the study, up to their hospital or NICU discharge.
Groups:
- Warming Mattress and Sterile Polyethylene Wrap Group-Mothers; Warming Mattress and Sterile Polyethylene Wrap Group-Infants: In the intervention group, the infant will be placed on the thermal mattress, then wrapped.
  Neonatal warming mattress: Babies will be warmed with a standard neonatal transport warming mattress immediately after birth.
  Sterile polyethylene wrap: Babies will be wrapped in a sterile polyethylene wrap prior to arrival at the warmer.
- Standard of Care Group-Mothers; Standard of Care Group-Infants: In the non-intervention group, the infant will be delivered onto the sterile field as per standard of care.
Arm/Group | Warming Mattress and Sterile Polyethylene Wrap Group-Mothers | Standard of Care Group-Mothers | Warming Mattress and Sterile Polyethylene Wrap Group-Infants | Standard of Care Group-Infants
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 1/25 | 1/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 2/25 | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Warming Mattress and Sterile Polyethylene Wrap Group-Mothers (N=25) | Standard of Care Group-Mothers (N=25) | Warming Mattress and Sterile Polyethylene Wrap Group-Infants (N=25) | Standard of Care Group-Infants (N=25)
Elevated temperature (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT04827394/Prot_SAP_000.pdf